CLINICAL TRIAL: NCT04009187
Title: Efficacy of a Wheelchair Propulsion Training Program for Manual Wheelchair Users: a Pilot Study
Brief Title: A Wheelchair Propulsion Training Program
Acronym: HS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Kerri Morgan, Assistant Professor of Occupational Therapy and Neurology, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201711056
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2020-04

CONDITIONS: Spinal Cord Injuries; Multiple Sclerosis; Amputation; Spina Bifida
Keywords: manual wheelchair; wheelchair propulsion; motor learning
MeSH Terms: conditions — Spinal Cord Injuries; Multiple Sclerosis; Spinal Dysraphism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Training group (Active Comparator): Training group will first receive 30 minutes of education about biomechanically efficient propulsion techniques. They will be tested on this knowledge to make sure participants understand the material. The participant then will be asked to come into the lab for 6 sessions of training, two times per week for three weeks. The training is an hour of the proper wheelchair propulsion techniques broken into 5 parts, 7 minutes each with breaks. Based on the motor learning principles, we gradually increase the components of the training by focusing either hand reaching toward the back of the wheel or hands reaching down toward the axle.
  Interventions: Behavioral: In-person wheelchair propulsion training program; Behavioral: 30-minute education session
- Control group (Active Comparator): Control group will first receive 30 minutes of education about the biomechanically efficient propulsion. They will be tested on this knowledge to make sure participants understand the material. No further training will be implemented with this group.
  Interventions: Behavioral: 30-minute education session

INTERVENTIONS:
Behavioral: In-person wheelchair propulsion training program — The wheelchair propulsion (WP) intervention is based on our previous pilot work and the best available evidence on WP training. The CPGs recommend minimizing the force and frequency of pushes while using long strokes during propulsion. Each training session will include massed practice with repetitions overground. Each session is organized to limit the number of variables (i.e., long push strokes and dropping the hands down below axle) presented to the participant at one time. Propulsion Set A will focus on using longer push strokes. Propulsion Set B will focus on dropping the hand down toward the axle. Propulsion Set C will focus on both A and B.
  Arms: Training group
Behavioral: 30-minute education session — Both groups will receive a 30-minute education session regarding the CPGs. This education session will follow the instructions provided in Rice and colleagues. (L. A. Rice et al., 2014). It consists of the importance of practicing biomechanical efficient propulsion. The material lists out the consequences and the impact of upper limb pain and injury. It provides a detailed step by step on how to propel properly. They will view the video that shows the biomechanics of efficient and inefficient propulsion.

SUMMARY:
The overall purpose of this project is to test the feasibility of a manual wheelchair propulsion program which aims to reduce the chance of development of upper limbs pain and injury.

DETAILED DESCRIPTION:
The purpose of this project is to develop a feasible wheelchair propulsion training that can fit into an in-patient rehabilitation schedule, and determine the effectiveness of the training protocol. This project consists of a randomized control trial (RCT) for manual wheelchair users (MWUs) that examines the number of manual wheelchair propulsion repetitions required to produce change. For the RCT, we will recruit twenty individuals who use manual wheelchairs as their primary means of mobility and who do not follow the recommended clinical guidelines for propulsion. Participants will be randomized into two independent groups: motor learning repetitions overground (Training Group; n =10), and general education on recommended propulsion techniques (Education Group; n =10). Demographics, cognition, shoulder strength, participation, and wheelchair seating may only be assessed at baseline. Participants then may be assessed from the kinematics of their wheelchair performance overground and on a motorized treadmill. Participants may be tested on their wheelchair propulsion techniques in and outside of the lab, upper extremity pain at baseline, post-intervention, and three-week follow-up; participants may also be asked qualitative questions regarding the intervention experience, the experience with the equipment and the laboratory research, the monitoring setting, and the general experience with the research study.

The primary research question is that will repetition of proper propulsion technique practiced overground result in improved manual wheelchair propulsion biomechanics?

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* have a mobility limitation requiring the use of a manual wheelchair (MWC)
* be able to self-propel a MWC bilaterally with their upper extremities
* plan to use a MWC for at least 75% of their activities throughout the day
* live in the community
* understand English at a sixth-grade level or higher
* can follow multi-step instructions
* able to provide informed consent independently
* able to tolerate propelling their wheelchair independently for 10m
* be willing to participate in three assessments and six training sessions at the Enabling Mobility in the Community Laboratory (EMC Lab).

Exclusion Criteria:

* maneuver their MWC with their lower extremities or with only one upper extremity
* display the proper wheelchair propulsion techniques during the screening process
* MWC position inhibits them from following the CPGs
* bilateral incoordination
* upper extremity strength inequalities resulting in a 12-inch deviation from a marked pathway
* surgeries compromising the integrity of the upper extremities
* cardiovascular complications within the past year
* upper extremity or overall bodily pain is rated 8/10 or higher per the Wong-Baker FACES Numeric Pain Scale (FACES)
* currently receiving medical treatment for an acute upper extremity injury
* have a Stage IV pressure injury or are currently hospitalized

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2019-10-22 (Actual); Study Completion 2019-10-22 (Actual)

PRIMARY OUTCOMES:
Motion capture - changes in push angle | Baseline, 3-week after baseline for the control group/immediate after training group intervention, 3-weeks after second assessment
  Push angle during the push phase of propulsion is assessed with video motion capture (VMC). The VMC system consists of 14 Vero 2.2 digital cameras to detect the location of the reflective markers, specifically on the shoulder, elbow, and wrist. The 3D infrared coordinates will be recorded while participants propel their wheelchair over the ground and on a dynamic roller system. Push angle will be calculated by finding the inner product of the vectors formed by the elbow-shoulder and elbow-wrist. The push angles will be compared across the three testing sessions. This variable corresponds to the recommendations outlined in the clinical practice guidelines. We hypothesize that the increase of push angle will be greater in the training group than the control group.
Motion capture - changes in hand-axle distance | Baseline, 3-week after baseline for the control group/immediate after training group intervention, 3-weeks after second assessment
  Hand-axle distance during the recovery phase of propulsion assessed with video motion capture (VMC). The VMC system consists of 14 Vero 2.2 digital cameras to detect the location of the reflective markers, specifically on the axle and the third metacarpal joint. The 3D infrared coordinates will be recorded while participants propel their wheelchair over the ground and on a dynamic roller system. Hand-axle distance will be calculated by the magnitude of the vector formed by the third metacarpal joint and the axle. The hand-axle will be compared across the three testing sessions. This variable corresponds to the recommendations outlined in the clinical practice guidelines. We hypothesize that the increase of hand-axle distance will be greater in the training group than the control group.
Wheelchair Propulsion Test (WPT) - changes in effectiveness | Baseline, 3-week after baseline for the control group/immediate after training group intervention, 3-weeks after second assessment
  The WPT assesses wheelchair mobility and performance of manual wheelchair users (MWU). The WPT requires MWU to propel using a self-selected natural velocity across 10 meters of a smooth flat surface from a static start. The number of pushes and the time will be recorded. The effectiveness of the propulsion is the displacement per push and will be calculated by the 10 meters divided by the number of pushes. We hypothesize that the increase in the effectiveness of propulsion will be greater in the training group than the control group.
Wheelchair Propulsion Test (WPT) - changes in cadence | Baseline, 3-week after baseline for the control group/immediate after training group intervention, 3-weeks after second assessment
  The WPT assesses wheelchair mobility and performance of manual wheelchair users (MWU). The WPT requires MWU to propel using a self-selected natural velocity across 10 meters of a smooth flat surface from a static start. The number of pushes and the time will be recorded. The cadence of the propulsion is the number of push per second and will be calculated by the number of push divided by the time spent finishing the 10-meters line. We hypothesize that the decrease of cadence will be greater in the training group than the control group.
Wheelchair Propulsion Test (WPT) - changes in propulsion pattern | Baseline, 3-week after baseline for the control group/immediate after training group intervention, 3-weeks after second assessment
  The WPT assesses wheelchair mobility and performance of manual wheelchair users (MWU). The WPT requires MWU to propel using a self-selected natural velocity across 10 meters of a smooth flat surface from a static start. The number of pushes and the time will be recorded. Clinicians will also record whether"during the contact phases, did the subject generally begin the contact between the hands and the hand-rims behind the top dead center of the rear wheel?", and " during the recovery phases, did the subject generally use a path of the hands that was predominantly beneath the handrims?" The clinician will provide his/her evaluation by answering the two questions. It is expected that after the training, the subject will change his/her pattern from both "no" to both "yes". These two questions are based on the clinical practice guidelines (CPG) and only when both answers are "yes", then the participant will be considered following CPG.
Outdoor propulsion - ratio of efficient propulsion pattern | Baseline, 3-week after baseline for the control group/immediate after training group intervention, 3-weeks after second assessment
  During the outdoor propulsion session, participants will push their wheelchair in an outdoor, asphalt surface parking lot with no ceiling for approximately three to five minutes across approximately 200 meters. The parking lot consists of 5°-10°slopes, a flat surface with small potholes, and two small bumps/thresholds. Participants will be told to propel their wheelchair at their regular speed in the parking lot. An experimenter will follow the participant with a body harnessed action camera to record participant's left side propulsion. A video coder will be viewing the recording then judge whether each push with the two questions mentioned in WPT form. The changes in propulsion patterns will be calculated by the amount of CPG-based propulsion divided by the total amount of propulsion. We hypothesize that the ratio increases of the CPG-based propulsion will be greater in the training group than controls.

CONTACTS AND LOCATIONS:
Overall Officials: Kerri Morgan, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Boninger ML, Souza AL, Cooper RA, Fitzgerald SG, Koontz AM, Fay BT. Propulsion patterns and pushrim biomechanics in manual wheelchair propulsion. Arch Phys Med Rehabil. 2002 May;83(5):718-23. doi: 10.1053/apmr.2002.32455. PMID 11994814
- [Background] Morgan KA, Tucker SM, Klaesner JW, Engsberg JR. A motor learning approach to training wheelchair propulsion biomechanics for new manual wheelchair users: A pilot study. J Spinal Cord Med. 2017 May;40(3):304-315. doi: 10.1080/10790268.2015.1120408. Epub 2015 Dec 16. PMID 26674751
- [Background] Will, K., Engsberg, J. R., Foreman, M., Klaesner, J., Birkenmeier, R., & Morgan, K. A. (2015). Repetition based training for efficient propulsion in new manual wheelchair users. Journal of Physical Medicine, Rehabilitation & Disabilities, 1(001), 1-9.
- [Background] Morgan KA, Engsberg JR, Gray DB. Important wheelchair skills for new manual wheelchair users: health care professional and wheelchair user perspectives. Disabil Rehabil Assist Technol. 2017 Jan;12(1):28-38. doi: 10.3109/17483107.2015.1063015. Epub 2015 Jul 3. PMID 26138222
- [Background] Paralyzed Veterans of America Consortium for Spinal Cord Medicine. Preservation of upper limb function following spinal cord injury: a clinical practice guideline for health-care professionals. J Spinal Cord Med. 2005;28(5):434-70. doi: 10.1080/10790268.2005.11753844. No abstract available. PMID 16869091
- [Background] Sawatzky B, DiGiovine C, Berner T, Roesler T, Katte L. The need for updated clinical practice guidelines for preservation of upper extremities in manual wheelchair users: a position paper. Am J Phys Med Rehabil. 2015 Apr;94(4):313-24. doi: 10.1097/PHM.0000000000000203. PMID 25299526
- [Background] Askari S, Kirby RL, Parker K, Thompson K, O'Neill J. Wheelchair propulsion test: development and measurement properties of a new test for manual wheelchair users. Arch Phys Med Rehabil. 2013 Sep;94(9):1690-8. doi: 10.1016/j.apmr.2013.03.002. Epub 2013 Mar 14. PMID 23499781
- [Background] MacPhee AH, Kirby RL, Coolen AL, Smith C, MacLeod DA, Dupuis DJ. Wheelchair skills training program: A randomized clinical trial of wheelchair users undergoing initial rehabilitation. Arch Phys Med Rehabil. 2004 Jan;85(1):41-50. doi: 10.1016/s0003-9993(03)00364-2. PMID 14970966
- [Background] Axelson, P., Chesney, D. Y., Minkel, J., & Perr, A. (1996). The manual wheelchair training guide. Santa Cruz, CA: Pax Press,1996.
- [Background] Kirby RL, Dupuis DJ, Macphee AH, Coolen AL, Smith C, Best KL, Newton AM, Mountain AD, Macleod DA, Bonaparte JP. The wheelchair skills test (version 2.4): measurement properties. Arch Phys Med Rehabil. 2004 May;85(5):794-804. doi: 10.1016/j.apmr.2003.07.007. PMID 15129405
- [Background] Rice IM, Pohlig RT, Gallagher JD, Boninger ML. Handrim wheelchair propulsion training effect on overground propulsion using biomechanical real-time visual feedback. Arch Phys Med Rehabil. 2013 Feb;94(2):256-63. doi: 10.1016/j.apmr.2012.09.014. Epub 2012 Sep 26. PMID 23022092
- [Background] DeGroot KK, Hollingsworth HH, Morgan KA, Morris CL, Gray DB. The influence of verbal training and visual feedback on manual wheelchair propulsion. Disabil Rehabil Assist Technol. 2009 Mar;4(2):86-94. doi: 10.1080/17483100802613685. PMID 19253097
- [Background] Rice LA, Smith I, Kelleher AR, Greenwald K, Boninger ML. Impact of a wheelchair education protocol based on practice guidelines for preservation of upper-limb function: a randomized trial. Arch Phys Med Rehabil. 2014 Jan;95(1):10-19.e11. doi: 10.1016/j.apmr.2013.06.028. Epub 2013 Jul 13. PMID 23856151
- [Background] Klaesner J, Morgan KA, Gray DB. The development of an instrumented wheelchair propulsion testing and training device. Assist Technol. 2014 Spring;26(1):24-32. doi: 10.1080/10400435.2013.792020. PMID 24800451